CLINICAL TRIAL: NCT02720133
Title: Ramadan Fasting Effects in Patients With Cardiovascular Risk Factors
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Head of departement, University of Monastir
Other Study IDs: GR2
Record Dates: First submitted 2014-07-24; First posted 2016-03-25 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Cardiovascular Risk Factors; Fasting
Keywords: ramadan fasting; variation of biochemical parameters; variation of hematological parameters; verify now assay
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with cardiovascular risk factors who fast Ramadan: Stable clinical and biochemical parameters before Ramadan fasting
  Interventions: Biological: biochemical parameters

INTERVENTIONS:
Biological: biochemical parameters — patients will be collected for analysis of blood standard examinations such as blood glucose, electrolytes (potassium, sodium, magnesium calcium), renal function and also the blood count, platelet aggregation.
  All these tests should be practice before, during and after Ramadan fasting for comparison.
  Other Names: hematological parameters assay; verify now assay

SUMMARY:
Ramadan Fasting has multiple effects on the variation of hematological and biochemical parameters.

DETAILED DESCRIPTION:
This is a prospective observational study, including patients with cardiovascular risk factors and doing the fast of Ramadan with assessment before, during and after the month of Ramadan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cardiovascular risk factors in stable conditions
* Ramadan fasting

Exclusion Criteria:

* Impossibility, contraindication or interruption of fasting

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stable patients with cardiovascular risk factors who fast during Ramadan
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
all cause clinical complications | 5 years

SECONDARY OUTCOMES:
evidence of acute coronary complications | 5 years

OTHER OUTCOMES:
clopidogrel and aspirin related complications | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, Pr., Principal Investigator — University Hospital Of Monastir Tunisia
Locations (1):
- Emergency Departement, Monastir, Non-US/Canada, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Attarzadeh Hosseini SR, Hejazi K. The effects of ramadan fasting and physical activity on blood hematological-biochemical parameters. Iran J Basic Med Sci. 2013 Jul;16(7):845-9. PMID 23997915
- [Derived] Bouida W, Beltaief K, Baccouche H, Sassi M, Dridi Z, Trabelsi I, Laaouiti K, Chakroun T, Hellara I, Boukef R, Sakly N, Hassine M, Added F, Razgallah R, Najjar F, Nouira S; Ramadan Research Group. Effects of Ramadan fasting on aspirin resistance in type 2 diabetic patients. PLoS One. 2018 Mar 12;13(3):e0192590. doi: 10.1371/journal.pone.0192590. eCollection 2018. PMID 29529091
- [Derived] Bouida W, Baccouche H, Sassi M, Dridi Z, Chakroun T, Hellara I, Boukef R, Hassine M, Added F, Razgallah R, Khochtali I, Nouira S; Ramadan Research Group. Effects of Ramadan fasting on platelet reactivity in diabetic patients treated with clopidogrel. Thromb J. 2017 Jun 2;15:15. doi: 10.1186/s12959-017-0138-0. eCollection 2017. PMID 28588426
- See also: The effects of ramadan fasting and physical activity on glycemic control, lipid metabolism, and the effects clopidogrel and aspirin activityameters. — http://www.ncbi.nlm.nih.gov/pubmed/23997915